CLINICAL TRIAL: NCT07075146
Title: Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate COmpared With Bictegravir/Emtricitabine/Tenofovir Alafenamide in ART-Naïve People Living With HIV and Overweight or Obesity
Brief Title: DOR/TDF/3TC COmpared With BIC/FTC/TAF in ART-Naïve People Living With HIV and Overweight or Obesity
Acronym: COATL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: José Antonio Mata Marín (Other Government)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Sponsor-Investigator, José Antonio Mata Marín, Principal investigator, Instituto Mexicano del Seguro Social
Organization: Instituto Mexicano del Seguro Social (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2025-3502-101
Record Dates: First submitted 2025-06-28; First posted 2025-07-20 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: HIV - Human Immunodeficiency Virus; Obesity; Overweight and/or Obesity
Keywords: HIV; overweight; obesity; Doravirine; Bictegravir
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: Study design: Experimental, longitudinal, prospective, randomized 1:1, open-label.
  Study type: Open-label, randomized clinical trial. Study location: Infectious Diseases Hospital. Study duration: 144 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIC/TAF/FTC (Active Comparator): Bictegravir/ tenofovir alafenamide/ emtricitabine 50/ 25/ 200 mg. It is the usual therapy, consisting of 3 drugs in a single tablet, based on an integrase inhibitor, and 2 nucleoside analogues, it is the experimental group
  Interventions: Drug: BIC/FTC/TAF
- DOR/3TC/TDF (Experimental): Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate 100/300/300 mg Non-nucleoside reverse transcriptase inhibitor (doravirine) Nucleoside reverse transcriptase inhibitors (lamivudine, tenofovir disoproxil fumarate)
  Interventions: Drug: DOR/3TC/TDF

INTERVENTIONS:
Drug: DOR/3TC/TDF — It is a triple-drug antiretroviral drug co-formulated in a single tablet. It contains Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate 100/300/300 mg
  Arms: DOR/3TC/TDF
Drug: BIC/FTC/TAF — It is a triple-drug antiretroviral drug co-formulated in a single tablet. It contains bictegravir 50 mg, tenofovir alafenamide 25 mg, and emtricitabine 200 mg. It is the standard therapy.
  Arms: BIC/TAF/FTC

SUMMARY:
Background:Historically, HIV infection was associated with significant weight loss. However, weight gain is now commonly observed after initiating antiretroviral therapy (ART), particularly in individuals underweight at baseline. It remains unclear whether this weight gain reflects a "return to health" or results from drug-related or metabolic effects, and whether it persists beyond immune restoration. Recent evidence indicates that ART regimens containing second-generation integrase strand transfer inhibitors (INSTIs), such as bictegravir combined with tenofovir alafenamide, are associated with greater weight gain compared to other antiretroviral combinations, raising concerns about potential long-term metabolic consequences.Objective:To evaluate the effectiveness, safety, and tolerability of Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate (DOR/3TC/TDF) compared with Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/FTC/TAF) in ART-naïve people living with HIV (PWH) who are overweight or obese.Materials and Methods:This open-label, randomized clinical trial, approved by the Ethics and Scientific Research Committee (No. 3502), will be conducted at the Infectious Diseases Hospital of the National Medical Center "La Raza" from May 2025 to May 2027. ART-naïve PWH, recently diagnosed, with no prior use of pre-exposure prophylaxis (PrEP) or post-exposure prophylaxis (PEP), who do not require hospitalization, and have a body mass index (BMI) ≥25 kg/m² and body fat >20%, will be invited to participate. Participants will provide written informed consent and be randomized 1:1 to receive either DOR/3TC/TDF or BIC/FTC/TAF.

DETAILED DESCRIPTION:
Study Assessments Measurements: Laboratory tests, vital signs, and body composition (via bioimpedance) will be assessed at weeks 4, 12, 24, 36, 48, 72, 96, 120, and 144. HIV viral load and CD4+ count will be measured at weeks 12, 24, 48, 72, 96, 120, and 144.Statistical Methods: Non-probabilistic sampling will be used. Data distribution will be evaluated with the Kolmogorov-Smirnov test. Descriptive statistics (means, medians, percentages) will be reported. Between-group comparisons will use the Mann-Whitney U test for continuous variables and chi-square or Fisher's exact test for categorical variables. Longitudinal analysis at weeks 12, 24, 48, 96, and 144 will employ the Wilcoxon test. A p-value ≤0.05 with a 95% confidence interval will indicate statistical significance.Study ProcedureEligible ART-naïve PWH attending the HIV clinic will be identified and invited to participate. After providing informed consent, participants will be informed that participation is voluntary and can be withdrawn at any time without consequences.

Baseline Visit

* Data Collection: A medical interview will gather sociodemographic, clinical, and comorbidity data, as well as lifestyle habits (diet, physical activity, alcohol use, smoking).
* Anthropometric Measurements: Conducted using a 4-point segmental bioimpedance scale (FitScan Segmental Body Composition Monitor C-545F) to assess weight, water percentage, muscle mass, bone mass, and fat percentage. Waist and hip circumference, blood pressure, heart rate, respiratory rate, and oxygen saturation will also be measured.
* Laboratory Assessments: Include glucose, creatinine, cystatin C, serum and urinary electrolytes, lipid profile, liver function tests, elastography (visceral and subcutaneous fat), complete blood count, HIV viral load, CD4+ count, hepatitis B and C serologies, and VDRL.

Randomization and Follow-Up Participants will be randomized using the MEDSHARING digital system to either DOR/3TC/TDF or BIC/FTC/TAF. Follow-up visits will occur at specified intervals through week 144. Adverse events will be monitored using the DAIDS grading scale. Neuropsychiatric assessments will use the Hospital Anxiety and Depression Scale (HADS), Insomnia Severity Index (ISI), and Patient Health Questionnaire (PHQ-9). Treatment satisfaction and distress will be evaluated with the HIV Treatment Satisfaction Questionnaire (HIVTSQ) and HIV Symptom Distress Module (HIVSDM).

Sampling and Sample Size

Simple random sampling will be employed. The sample size is 306 participants per group, calculated based on:

* 80% statistical power
* Alpha level of 0.05
* 12% non-inferiority margin
* 80% expected virologic response at week 48
* 10% attrition rate Statistical Analysis
* Categorical Variables: Reported as frequencies and percentages.
* Continuous Variables: Described using means ± standard deviations or medians with interquartile ranges.
* Statistical Tests:

  * Between-group comparisons: Mann-Whitney U or Student's t-test
  * Within-group comparisons: Wilcoxon or paired t-test
  * Multiple time points: Friedman or repeated-measures ANOVA
  * Associations: Chi-square or Fisher's exact test
  * Multivariate analysis: Binary logistic regression
* Software: SPSS v29.0.2 for Mac (IBM) will be used for data analysis. Ethical Considerations and Data Confidentiality The study adheres to the Declaration of Helsinki, CIOMS/WHO, and ICH-GCP guidelines. Approval has been obtained from the institutional Ethics and Research Committee. Participant confidentiality will comply with IMSS policy and Mexican regulations, using anonymized unique codes. Only standard-of-care treatments per national and international guidelines will be used. Risks are minimal, primarily related to venipuncture, with medical evaluation and treatment provided as needed

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years) with confirmed HIV diagnosis, ART-naïve
2. Signed informed consent
3. HIV-1 RNA ≥1000 copies/mL
4. No history of PrEP or PEP failure
5. BMI ≥25 kg/m² and body fat >20%
6. Stable treatment for dyslipidemia (if applicable)
7. No planned medication changes affecting weight
8. Willingness to adhere to assigned ART
9. Recent HIV-1 RNA and CD4+ results
10. GFR (CKD-EPItip) ≥60 mL/min
11. ALT and AST <90 IU/L
12. Willingness to report dietary or physical activity changes during follow-up Non-Inclusion Criteria

1. Uncontrolled diabetes 2. Recent changes in insulin or hypoglycemic drugs (<3 months) 3. Active malignancy 4. History of bariatric surgery 5. Allergies to study drugs 6. Hepatitis B and/or C coinfection 7. GFR <60 mL/min (CKD-EPI) 8. Drug interactions with ART regimens 9. Recent (60 days) use of anorectic drugs 10. Recent (30 days) hospitalization for severe illness 11. Unstable hypothyroidism

Exclusion Criteria:

1. Loss of social security coverage
2. Newly discovered allergy to study drugs
3. Withdrawal of consent
4. Hepatitis B or C infection acquired during follow-up
5. Use of psychiatric or thyroid medications without a stable dose for ≥12 weeks
6. Initiation or discontinuation of medications affecting weight after enrollment
7. Unplanned bariatric surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
To determine the safety and tolerability of Doravirine/Lamivudine/Tenofovir compared with Bictegravir/Tenofovir Alafenamide/Emtricitabine in ART-naive people living with HIV at 144 weeks of treatment. | 144 weeks
  Number of participants with treatment-related adverse events as assessed of serious adverse events (WHO grade 3 or 4) for PWH treated with DOR/TDF/3TC or BIC/FTC/TAF at 144 weeks, expressed in proportions of new cases.
Evaluate the effectiveness and safety of Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate (DOR/3TC/TDF) compared with Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/FTC/TAF) | 144 weeks of follow-up with interim analysis at 48 and 96 weeks
  Effectiveness: Number of participants with viral load measurement (HIV-1 RNA) <50 copies/mL at 144 weeks of follow-up for PWH treated with DOR/3TC/TDF or BIC/FTC/TAF,BIC/FTC/TAF at 144 weeks,

SECONDARY OUTCOMES:
To compare changes in lipid profile in people living with HIV (PLWH) treated with Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate versus Bictegravir/Emtricitabine/Tenofovir Alafenamide after initiating ART | 144 weeks, with interim analyses at 24,48,72, 96 , 120, and 144 weeks
To compare changes in body composition in PLWH treated with Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate versus Bictegravir/Emtricitabine/Tenofovir Alafenamide before initiating ART | 144 weeks, with interim analyses at 24,48,72, 96 , 120, and 144 weeks
  Changes of percentage of fat
To compare changes in estimated glomerular filtration rate (eGFR) in PLWH treated with Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate versus Bictegravir/Emtricitabine/Tenofovir Alafenamide after initiating TAR | 144 weeks, with interim analyses at 24,48,72, 96 , 120, and 144 weeks
  To compare changes in kidney function using cystatin C and creatinine levels calculated using the 2021 CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) equation: Creatinine-Cystatin C expressed in ml/min/1.73 m2.
  Classifying kidney function stages:
  Stage 1: Normal (GFR >90 ml/min/m2) Stage 2: Mild (GFR 60-89 ml/min/m2) Stage 3: Moderate (GFR 30-59 ml/min/m2) Stage 4: Severe (GFR 15-29 ml/min/m2) Stage 5: Renal failure for dialysis (GFR <15 ml/min/m2)
To compare changes in cardiovascular risk using the Framingham Risk Score and the Pooled Cohort Equations (ASCVD AHA/ACC) in PLWH treated with Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate versus Bictegravir/Emtricitabine/Tenofovir Alafenamide | 144 weeks, with interim analyses at 24,48,72, 96 , 120, and 144 weeks
  To evaluate and compare changes in cardiovascular risk based on the ASCVD (Atherosclerotic Cardiovascular Disease) 2013 Risk Calculator from American College of Cardiology (ACC) and American Heart Association in ART-naive PWH initiating DOR/3TC/TDF regimen compared with BIC/FTC/TAF after 144 weeks of follow-up.
  To evaluate in percentages of risk High cardiovascular risk: ≥20% Borderline cardiovascular risk: ≥5%-<7.5% Low cardiovascular risk: <5% The score is directly proportional to the risk, and determines the 10-year risk of ASCVD, (Atherosclerotic Cardiovascular Disease) for example: myocardial infarction, stroke, or death due to coronary heart disease or stroke

CONTACTS AND LOCATIONS:
Overall Officials: José A Mata, M.Sc, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Hospital de infectología, Centro Médico Nacional La Raza, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
Participant data are confidential and may be requested from the principal investigator.

REFERENCES:
- [Background] Kousari AE, Wilson MP, Hawkins KL, Bandali MM, Henao-Martinez AF, Gardner EM, Erlandson KM. Weight change with antiretroviral switch from integrase inhibitor or tenofovir alafenamide-based to Doravirine-Based regimens in people with HIV. HIV Res Clin Pract. 2024 Dec;25(1):2339576. Epub 2024 Jun 3. PMID 38831550
- [Background] Orkin C, Molina JM, Cahn P, Lombaard J, Supparatpinyo K, Kumar S, Campbell H, Wan H, Teal V, Jin Xu Z, Asante-Appiah E, Sklar P, Teppler H, Lahoulou R; DRIVE-FORWARD and DRIVE-AHEAD collaborators. Safety and efficacy of doravirine as first-line therapy in adults with HIV-1: week 192 results from the open-label extensions of the DRIVE-FORWARD and DRIVE-AHEAD phase 3 trials. Lancet HIV. 2024 Feb;11(2):e75-e85. doi: 10.1016/S2352-3018(23)00258-8. Epub 2023 Dec 20. PMID 38141637